CLINICAL TRIAL: NCT06303492
Title: Aspiration Risk Assessment by Gastric Ultrasound in eMErgency Surgery and ANesThetic Decision-making: a Multicentre Mixed Method Study- The ARGUMENT Study
Brief Title: Aspiration Risk Assessment by Gastric Ultrasound in eMErgency Surgery and ANesThetic Decision-making: The ARGUMENT Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: CTO 4096
Record Dates: First submitted 2024-02-28; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-02

CONDITIONS: Pulmonary Aspiration; Emergency Surgery

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gastric ultrasound (GUS) group (Experimental): Aspiration risk assessment using GUS in addition to the standard clinical assessment.
  Interventions: Procedure: GUS
- Control (No Intervention): Aspiration risk assessment only by standard clinical assessment, and no GUS

INTERVENTIONS:
Procedure: GUS — Aspiration risk assessment by GUS
  Arms: Gastric ultrasound (GUS) group

SUMMARY:
Pulmonary aspiration of gastric contents is a serious patient safety problem accounting for 50% of anesthesia-related mortality. The risk is higher in patients undergoing emergency surgery as the gastric content is uncertain which poses a challenge to anesthetic decision-making. Standard clinical assessment to identify at-risk patients primarily relies on preoperative fasting guidelines and is not adequate for patients undergoing emergency surgeries. Point-of-care gastric ultrasound (GUS) has emerged as an accurate bedside tool providing information regarding the type and volume of gastric contents. When GUS was added to standard clinical assessment, anesthetic management plan changed in 71% of adult elective and 37% of pediatric emergency surgical procedures. Such data is lacking in adult patients undergoing emergency surgeries. The investigators propose a multicentre mixed-method study to evaluate the impact of GUS on aspiration risk assessment and subsequent Anesthetic Plan before emergency surgeries. The evidence from this study will improve patient safety by accurately identifying patients at risk of aspiration and tailoring anesthetic techniques and airway management to prevent pulmonary aspiration in patients undergoing emergency surgeries.

DETAILED DESCRIPTION:
The proposed trial design is a mixed-method, multicenter study that includes a randomized controlled trial (RCT) and a qualitative assessment component. The RCT will evaluate the impact of adding GUS to the standard clinical assessment on the incidence of changes in the anesthetic plan for adult patients undergoing emergency surgery. The qualitative assessment will gather attending anesthesiologists' opinions on the addition of GUS in an emergency surgical setting.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* American Society of Anesthesiologists' (ASA) physical status I-III
* Patients scheduled for non-elective non-cardiac surgery.

Exclusion Criteria:

* Abnormal anatomy of the upper gastro-intestinal tract (including hiatus hernia, gastric tumors, and previous surgeries of the upper gastrointestinal tract).
* Extrinsic gastric compression obtained from the medical history or during the actual ultrasound examination.
* Pregnancy.
* Attending anesthesiologist refusal to include the patient for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of change in Anesthetic Plan | Baseline
  The primary outcome of the study is a change from the initial anesthetic plan after viewing GUS results in the intervention group, and after being given the opportunity to revise the plan in the control group.

SECONDARY OUTCOMES:
Percentage change in the three-category risk assessment before and after GUS | Baseline
  The secondary aim is only related to the intervention group, (1) to compare the aspiration risk assessment categories between the standard clinical assessment and GUS examination

IPD SHARING:
Plan to Share IPD: No